CLINICAL TRIAL: NCT01223937
Title: A Multi-centre, Randomised, Double-blind, Placebo-controlled, Parallel-group Trial to Demonstrate the Efficacy and Safety of Desmopressin Orally Disintegrating Tablet for the Treatment of Nocturia in Adult Females
Brief Title: Investigation of the Superiority Effect of Desmopressin to Placebo in Terms of Night Voids Reduction in Nocturia Adult Female Patients
Acronym: COMFORT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FE992026 CS40
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Results first posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-09

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desmopressin 25 μg (Experimental): Participants took 1 orally disintegrating tablet of desmopressin 25 μg every night approximately 1 hour before bedtime for the entire duration of the 3-month treatment period.
  Interventions: Drug: Desmopressin
- Placebo (Placebo Comparator): Participants took 1 orally disintegrating tablet of placebo every night approximately 1 hour before bedtime for the entire duration of the 3-month treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desmopressin
  Other Names: FE992026; MINIRIN®; Nocturin®
  Arms: Desmopressin 25 μg
Drug: Placebo
  Arms: Placebo

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled, parallel-group trial to investigate the safety and efficacy of desmopressin oral melt tablets against placebo during 3 months of treatment in adult females with nocturia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to performance of any trial-related activity
* Female sex 18 years of age or older
* At least 2 voids every night in a consecutive 3-day period during the screening period

Exclusion Criteria:

1. Evidence of severe daytime voiding dysfunction defined as:

   * Urge urinary incontinence (more than 1 episode/day in the 3-day diary period)
   * Urgency (more than 1 episode/day in the 3-day diary period)
   * Frequency (more than 8 daytime voids/day in the 3-day diary period)
2. Interstitial cystitis
3. Urinary retention or a post void residual volume in excess of 150 mL as confirmed by bladder ultrasound performed after suspicion of urinary retention
4. Habitual or psychogenic polydipsia (fluid intake resulting in a urine production exceeding 40 mL/kg/24 hours)
5. Central or nephrogenic diabetes insipidus
6. Syndrome of inappropriate anti-diuretic hormone secretion
7. Current or a history of urologic malignancies e.g. bladder cancer
8. Genitourinary tract pathology e.g., infection or stone in the bladder and urethra causing symptoms
9. Neurogenic detrusor activity (detrusor overactivity).
10. Suspicion or evidence of cardiac failure
11. Uncontrolled hypertension
12. Uncontrolled diabetes mellitus
13. Hyponatraemia: Serum sodium level must be within normal limits
14. Renal insufficiency: Serum creatinine must be within normal limits and estimated glomerular filtration rate must be more than or equal to 50 mL/min
15. Hepatic and/or biliary diseases: Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) levels must not be more than twice the upper limit of normal range. Total bilirubin level must not be more than 1.5 mg/dL
16. History of obstructive sleep apnea
17. Previous desmopressin treatment for nocturia
18. Treatment with another investigational product within 3 months prior to screening
19. Concomitant treatment with any prohibited medication e.g., loop diuretics (furosemide, torsemide, ethacrynic acid) and any other investigational drug
20. Pregnancy, breastfeeding, or a plan to become pregnant during the period of the clinical trial. Subjects of reproductive age must have documentation of a reliable method of contraception. All pre-and perimenopausal subjects have to perform pregnancy tests. Amenorrhea of more than 12 months' duration based on the reported date of the last menstrual period is sufficient documentation of post-menopausal status and does not require a pregnancy test
21. Known alcohol or substance abuse
22. Work or lifestyle that may interfere with regular nighttime sleep e.g., shift workers
23. Any other medical condition, laboratory abnormality, psychiatric condition, mental incapacity, or language barrier that, in the judgment of the Investigator, would impair participation in the trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (45):
- United States (41):
  - Medical Affiliated Research Center Inc., Huntsville, Alabama
  - Radiant Research Inc., Scottsdale, Arkansas
  - Family Medical Center, Foothill Ranch, California
  - Axis Clinical Trials, Los Angeles, California
  - Radiant Research Inc., Santa Rosa, California
  - Downtown Woman's Health Care, Denver, Colorado
  - Front Range Clinical Research, Wheat Ridge, Colorado
  - South Florida Medical Research, Aventura, Florida
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - FPA Clinical Research, Kissimmee, Florida
  - Sunrise Medical Research, Lauderdale Lakes, Florida
  - DMI Research, Pinellas Park, Florida
  - Southeastern Institute, Columbus, Georgia
  - Southeastern Medical Research Institute, Columbus, Georgia
  - Radiant Research Inc., Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Accelovance, Peoria, Illinois
  - Accelovance, South Bend, Indiana
  - FutureCare Studies, Springfield, Massachusetts
  - Bay State Clinical Trials, Inc., Watertown, Massachusetts
  - Beyer Research, Paw Paw, Michigan
  - Remedica, LLC, Rochester, Michigan
  - Radiant Research, Inc., Edina, Minnesota
  - Radiant Research, Inc., St Louis, Missouri
  - Radiant Research, Las Vegas, Nevada
  - Anderson & Collins Clinical Research Inc, Edison, New Jersey
  - ACCUMED Research Associates, Garden City, New York
  - Center for Urologic Research of WNY, LLC, Williamsville, New York
  - Radiant Research, Inc., Akron, Ohio
  - Community Research, Cincinnati, Ohio
  - Complete HealthCare for Women, Columbus, Ohio
  - HWC Women's Research Center, Englewood, Ohio
  - Urologic Consultants of SE PA, Bala-Cynwyd, Pennsylvania
  - Philadelphia Clinical Research, LLC, Philadelphia, Pennsylvania
  - Radiant Research, Inc., Greer, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Radiant Research Inc., Dallas, Texas
  - Quality Research, Inc., San Antonio, Texas
  - Radiant Research, Inc., San Antonio, Texas
  - Exemplar Research Inc., Morgantown, West Virginia
- Canada (4):
  - CanMed Clinical Research Inc., Victoria, British Columbia
  - The Male/Female Health Research Center, Barrie, Ontario
  - Urology Associates/Urologic Medical Research, Kitchener, Ontario
  - Investigational site, North Bay, Ontario

REFERENCES:
- [Result] Sand PK, Dmochowski RR, Reddy J, van der Meulen EA. Efficacy and safety of low dose desmopressin orally disintegrating tablet in women with nocturia: results of a multicenter, randomized, double-blind, placebo controlled, parallel group study. J Urol. 2013 Sep;190(3):958-64. doi: 10.1016/j.juro.2013.02.037. Epub 2013 Feb 20. PMID 23454404
- [Derived] Juul KV, Malmberg A, van der Meulen E, Walle JV, Norgaard JP. Low-dose desmopressin combined with serum sodium monitoring can prevent clinically significant hyponatraemia in patients treated for nocturia. BJU Int. 2017 May;119(5):776-784. doi: 10.1111/bju.13718. Epub 2016 Dec 10. PMID 27862898

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization was stratified by age (<65 years, >= 65 years).
Period: Overall Study
Arm/Group | Placebo | Desmopressin 25 μg
Started | 131 (Intent to treat population: randomized participants regardless if they were exposed to treatment.) | 137 (Intent to treat population: randomized participants regardless if they were exposed to treatment.)
Full Analysis Set (FAS) | 128 (FAS: participants with at least one post-treatment efficacy assessment) | 133 (FAS: participants with at least one post-treatment efficacy assessment)
Safety Analysis Set (SAS) | 126 (SAS: participants with at least one post-treatment safety assessment) | 135 (SAS: participants with at least one post-treatment safety assessment)
Completed | 114 | 119
Not Completed | 17 | 18
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 1 | 4
Not completed — Adverse Event | 1 | 4
Not completed — Protocol Violation | 8 | 7
Not completed — Other | 4 | 1

BASELINE CHARACTERISTICS:
Population: Demographic data offered from the Full Analysis Set population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Desmopressin 25 μg | Total
Number analyzed (Participants) | 128 | 133 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (14.1) | 59.5 (14.3) | 59.8 (14.2)
Age, Customized [Number; unit: participants]
  < 65 years | 65 | 71 | 136
  >=65 years | 63 | 62 | 125
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 133 | 261
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 104 | 109 | 213
  Black/African American | 22 | 23 | 45
  Asian | 1 | 1 | 2
  Native Hawaiian/other Pacific Islander | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 17 | 26 | 43
  Not Hispanic or Latino | 111 | 107 | 218
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.1 (6.58) | 31.4 (7.03) | 30.3 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Number of Nocturnal Voids Averaged Over a 3-Month Period
Description: The number of nocturnal voids was the average over 3 consecutive 24-hour periods prior to Day 1 and prior to the during-treatment visits (Week 1, Months 1, 2, 3) as recorded in participant diaries. The first morning void was not counted as a nocturnal void. Change from baseline values for Week 1, and Months 1, 2 and 3 are reported below.
  Comparison of the mean number of nocturnal voids at baseline and over a 3-month treatment period (obtained by longitudinal analysis of Week 1, and Months 1, 2 and 3) are reported in the statistical analysis. This was the first co-primary endpoint. The trial was to be declared positive only if the 25 μg desmopressin group had a statistically significant positive effect as compared to placebo on both co-primary endpoints.
Time Frame: Day 1 (Baseline); Week 1, Months 1, 2, 3 (3-month treatment period)
Population: Full analysis set (FAS).
Measure: Mean (Standard Deviation); unit: nocturnal voids
Arm/Group | Placebo | Desmopressin 25 μg
Number analyzed (Participants) | 128 | 133
nocturnal voids
  Week 1 (n=124, 128) | -1 (0.94) | -1.21 (0.957)
  Month 1 (n=121, 126) | -1.25 (1.12) | -1.47 (1)
  Month 2 (n=116, 121) | -1.36 (1.12) | -1.57 (1.03)
  Month 3 (n=107, 113) | -1.38 (1.13) | -1.69 (0.978)
Statistical Analysis 1: Comparison: Placebo vs Desmopressin 25 μg; The trial was to be declared positive only if the 25 μg desmopressin group had a statistically significant positive effect as compared to placebo on both co-primary outcomes. A summary of mean change in nocturnal voids, assessed longitudinally during 3 months of treatment, is presented below for the FAS using LOCF; Test type: Superiority or Other; p = 0.0280, ANCOVA — A priori threshold for significance was p<=0.05; Repeated measures ANCOVA with treatment, visit (including a treatment-by-visit interaction term), and age stratification (<65, ≥65 years) as factors; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.42 to -0.02]

2. Primary Outcome: Adjusted Probability of Participants Achieving a >33% Reduction From Baseline in Number of Nocturnal Voids for All During-Treatment Visits up to Month 3
Description: Probability of participants achieving 33% responder status during 3 months of treatment employed a longitudinal analysis assessing nocturnal void information captured in the 3-day diary. A 33% responder was defined as a participant with a decrease of at least 33% in the mean number of nocturnal voids relative to baseline. The number of nocturnal voids was the average over 3 consecutive 24-hour periods prior to Day 1 and prior to the during treatment visits (Week 1, Months 1, 2, 3) as recorded in participant diaries. The first morning void was not counted as a nocturnal void.
  This was the second co-primary endpoint. The trial was to be declared positive only if the 25 μg desmopressin group had a statistically significant positive effect as compared to placebo on both co-primary endpoints.
Time Frame: Day 1 (Baseline); Week 1, Months 1, 2, 3 (3-month treatment period)
Population: Full analysis set (FAS).
Measure: Number; unit: probability
Arm/Group | Placebo | Desmopressin 25 μg
Number analyzed (Participants) | 128 | 133
probability | 0.64 | 0.76
Statistical Analysis 1: Comparison: Placebo vs Desmopressin 25 μg; The trial was to be declared positive only if the 25 μg desmopressin group had a statistically significant positive effect as compared to placebo on both co-primary outcomes; Test type: Superiority or Other; p = 0.0061, Generalized Estimating Equation (GEE) — A priori threshold for significance was p<=0.05; GEE Method with treatment, visit (including a treatment-by-visit interaction term), and age stratification (<65, ≥65 years) as factors; Odds Ratio (OR) = 1.85, 95% CI 2-sided [1.19 to 2.86]

3. Secondary Outcome: Change From Baseline in Mean Number of Nocturnal Voids at Month 3
Description: The number of nocturnal voids was the average over 3 consecutive 24-hour periods prior to Day 1 and prior to the during-treatment visits (Month 3 for this outcome) as recorded in participant diaries. The first morning void was not counted as a nocturnal void.
  Secondary efficacy outcomes (#3-7) used a hierarchical step-down approach in the order listed.
Time Frame: Day 1 (Baseline), Month 3
Population: Full Analysis Set (FAS), including participants with complete data supporting this outcome in the participant diary.
Measure: Mean (Standard Deviation); unit: nocturnal voids
Arm/Group | Placebo | Desmopressin 25 μg
Number analyzed (Participants) | 107 | 113
nocturnal voids | -1.38 (1.13) | -1.69 (0.978)
Statistical Analysis 1: Comparison: Placebo vs Desmopressin 25 μg; Change from baseline in the adjusted mean number of nocturnal voids in the FAS using LOCF; Test type: Superiority or Other; p = 0.0104, ANCOVA — A priori threshold for significance was p<=0.05; ANCOVA of change from baseline adjusted for age (<65, >=65) and baseline nocturnal voids, using last observation carried forward; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.54 to -0.07]

4. Secondary Outcome: Adjusted Probability of Participants Achieving a >33% Reduction From Baseline in Number of Nocturnal Voids at Month 3
Description: Probability of participants achieving 33% responder status at Month 3 employed a longitudinal analysis assessing nocturnal void information captured in the 3-day diary. A 33% responder was defined as a participant with a decrease of at least 33% in the mean number of nocturnal voids relative to baseline. The number of nocturnal voids was the average over 3 consecutive 24-hour periods prior to Day 1 and prior to the Month 3 visit as recorded in participant diaries. The first morning void was not counted as a nocturnal void.
  The secondary efficacy outcomes (#3-7) used a hierarchical step-down approach in the order listed.
Time Frame: Day 1 (Baseline), Month 3
Population: Full Analysis Set (FAS), including participants with complete data supporting this outcome in the participant diary.
Measure: Number; unit: probability
Arm/Group | Placebo | Desmopressin 25 μg
Number analyzed (Participants) | 107 | 113
probability | 0.69 | 0.79
Statistical Analysis 1: Comparison: Placebo vs Desmopressin 25 μg; Test type: Superiority or Other; p = 0.0586, Regression, Logistic — A priori threshold for significance was p<=0.05; Logistical regression of 33% responder status adjusted for age (<65, >=65) and baseline nocturnal voids using last observation carried forward; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.98 to 3.05]

5. Secondary Outcome: Change From Baseline in Mean Time to First Nocturnal Void at Month 3
Description: The time to first void was defined as the time from going to bed with the intention of sleeping until first nocturnal void or until waking in the morning in cases where there was no nocturnal void. The time to first void was derived from the sleep and voiding diary. The mean time to first void was calculated as the average over 3 consecutive 24-hour periods prior to the Month 3 visit.
  The secondary efficacy outcomes (#3-7) used a hierarchical step-down approach in the order listed.
Time Frame: Day 1 (Baseline), Month 3
Population: Full Analysis Set (FAS), including participants with complete data supporting this outcome in the participant diary.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Desmopressin 25 μg
Number analyzed (Participants) | 107 | 113
minutes | 115 (139) | 168 (138)
Statistical Analysis 1: Comparison: Placebo vs Desmopressin 25 μg; Test type: Superiority or Other; p = 0.0034, ANCOVA — A priori threshold for significance was p<=0.05; ANCOVA of change from baseline adjusted for age (<65, >=65) and baseline time to first nocturnal void, using last observation carried forward; Mean Difference (Final Values) = 49.03, 95% CI 2-sided [16.35 to 81.70]

6. Secondary Outcome: Change From Baseline in Nocturnal Urine Volume at Month 3
Description: The nocturnal urine volume was derived from the 3-day urine volume diary. The nocturnal urine volume included the volume of the first morning void. Mean urine volumes were calculated as the average over 3 consecutive 24-hour periods prior to the Month 3 visit.
  The secondary efficacy outcomes (#3-7) used a hierarchical step-down approach in the order listed.
Time Frame: Day 1 (Baseline), Month 3
Population: Full Analysis Set (FAS), including participants with complete data supporting this outcome in the participant diary.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Desmopressin 25 μg
Number analyzed (Participants) | 107 | 112
mL | -151 (262) | -242 (283)
Statistical Analysis 1: Comparison: Placebo vs Desmopressin 25 μg; Test type: Superiority or Other; p = 0.0031, ANCOVA — A priori threshold for significance was p<=0.05; ANCOVA of change from baseline adjusted for age (<65, >=65) and baseline nocturnal urine volume, using last observation carried forward; Mean Difference (Final Values) = -83.56, 95% CI 2-sided [-138.74 to -28.38]

7. Secondary Outcome: Change From Baseline in 24-Hour Urine Volume at Month 3
Description: Twenty-four hour urine volume was derived from the 3-day urine volume diary. Mean urine volumes were calculated as the average over 3 consecutive 24-hour periods prior to the Month 3 visit.
  The secondary efficacy outcomes (#3-7) used a hierarchical step-down approach in the order listed.
Time Frame: Day 1 (Baseline), Month 3
Population: Full Analysis Set (FAS), including participants with complete data supporting this outcome in the participant diary.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Desmopressin 25 μg
Number analyzed (Participants) | 101 | 111
mL | -152 (497) | -255 (522)
Statistical Analysis 1: Comparison: Placebo vs Desmopressin 25 μg; Test type: Superiority or Other; p = 0.1829, ANCOVA — A priori threshold for significance was p<=0.05; ANCOVA of change from baseline adjusted for age (<65, >=65) and baseline 24-hour urine volume, using last observation carried forward; Mean Difference (Final Values) = -72.91, 95% CI 2-sided [-180.42 to 34.60]

8. Secondary Outcome: Summary of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: A TEAE was any adverse event occurring after start of treatment and within the time of residual drug effect, i.e., within 1 day of the last dose of desmopressin. An adverse drug reaction (ADR) was any AE assessed by the Investigator as possibly/probably related to study drug.
Time Frame: Day 1 up to 3 months
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Desmopressin 25 μg
Number analyzed (Participants) | 126 | 135
participants
  All adverse events (AEs) | 57 | 60
  Severe AEs | 3 | 1
  Adverse drug reactions (ADRs) | 15 | 26
  AEs leading to discontinuation | 1 | 4
  ADRs leading to discontinuation | 0 | 3
  Serious AEs | 2 | 0
  Deaths | 0 | 0

9. Secondary Outcome: Minimum Post-Treatment Serum Sodium Levels
Description: Serum sodium levels were monitored since hyponatremia is a potential serious adverse event associated with daily doses of desmopressin. The serum sodium level must have been within the normal reference range at the Screening Visit for the participant to be eligible for enrollment. A participant was to be withdrawn from the trial if the serum sodium level was <=125 mmol/L at any time.
Time Frame: Day 1 up to 3 months
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Desmopressin 25 μg
Number analyzed (Participants) | 126 | 135
participants
  <=125 mmol/L | 0 | 0
  126-129 mmol/L | 0 | 3
  130-134 mmol/L | 2 | 11
  >=135 mmol/L | 124 | 121

ADVERSE EVENTS:
Time Frame: Day 1 up to 3 months
Arm/Group | Placebo | Desmopressin 25 μg
Serious Adverse Events (participants affected / at risk) | 2/126 | 0/135
Other Adverse Events (participants affected / at risk) | 14/126 | 12/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=126) | Desmopressin 25 μg (N=135)
Cellulitis (Infections and infestations) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=126) | Desmopressin 25 μg (N=135)
Headache (Nervous system disorders) | 4 (5) | 7 (7)
Urinary tract infection (Infections and infestations) | 10 (10) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.